CLINICAL TRIAL: NCT07125716
Title: Effects of Different Lengths of Surgical Sutures in Acupoint Catgut Implantation on Simple Abdominal Obesity in Adults
Brief Title: Suture Length Effects in Acupoint Implantation for Abdominal Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202500161A3
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Obesity; Obesity
MeSH Terms: conditions — Obesity, Abdominal; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 inch suture length (Experimental)
  Interventions: Device: 1 inch
- 0.5 inch suture length (Active Comparator)
  Interventions: Device: 0.5 inch

INTERVENTIONS:
Device: 1 inch — 1 inch suture length
  Arms: 1 inch suture length
Device: 0.5 inch — 0.5 inch suture length
  Arms: 0.5 inch suture length

SUMMARY:
Obesity is a metabolic disorder and has become a global health issue with a steadily increasing prevalence. According to the Health Promotion Administration's statistical report, the overweight and obesity rate among adults in Taiwan was 50.3% between 2017 and 2020. Based on the Ministry of Health and Welfare's criteria, a BMI ≥27 kg/m² is classified as obese.

Studies have shown that acupuncture can effectively reduce body weight with low cost and minimal side effects. Acupoint catgut embedding is a treatment method that combines traditional meridian acupuncture with modern medical materials by implanting surgical sutures into acupoints to provide continuous stimulation.

A 2022 systematic review found that catgut embedding is more effective than traditional acupuncture, requires fewer treatment sessions, and has a high safety profile. However, no studies have yet investigated whether different lengths of implanted surgical sutures affect treatment outcomes.

This study is a single-center, double-blind, randomized controlled trial aimed at identifying the optimal suture length for acupoint catgut embedding, in order to enhance its efficiency and therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign a written informed consent form
2. BMI ≥27 kg/m² (Ministry of Health and Welfare standard)
3. Waist circumference ≥90 cm for men
4. Waist circumference ≥80 cm for women
5. Age between 18 and 65 years

Exclusion Criteria:

1. Endocrine disorders (thyroid disease, pituitary disorders, and diabetes)
2. Autoimmune diseases (systemic lupus erythematosus, Sjögren's syndrome, and rheumatoid arthritis)
3. Heart diseases (heart failure, arrhythmia, etc.)
4. Abnormal liver function
5. Abnormal kidney function
6. Stroke within the past year
7. Pregnant or breastfeeding women
8. Coagulation disorders
9. Tumors
10. Participation in weight loss treatment within the past 6 months
11. Any other condition deemed unsuitable for the trial by the physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | 1 week,4 week,8 week

SECONDARY OUTCOMES:
hip circumference | 1 week,4 week,8 week
weight | 1 week,4 week,8 week
BMI | 1 week,4 week,8 week
VAS | 1 week,4 week,8 week
Ultrasound Fat Thickness | 1 week,4 week,8 week

CONTACTS AND LOCATIONS:
Locations (1):
- Chang-Geng Medical Foundation Keelung Chang-Geng Memorial Hospital, Keelung, Taiwan